CLINICAL TRIAL: NCT04614649
Title: Right Iliac Fossa Treatment-Turkey Audit
Acronym: RIFT-Turkey
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ali Yalcinkaya, Dr., Gazi University
Other Study IDs: RIFT-TR
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Abdominal Pain; Appendicitis; Appendicitis Acute
Keywords: appendicitis; appendectomy; right iliac fossa; abdominal pain
MeSH Terms: conditions — Abdominal Pain; Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Acute appendicitis stands out as a frequently encountered surgical emergency. Despite decades of experience and research, the diagnosis remains a formidable challenge, particularly in young females experiencing acute abdominal pain, where the assessment requires consideration of a broader spectrum of potential causes. An overarching concern lies in the risk of over-treatment, leading to an escalation in unnecessary surgeries, known as the negative appendectomy rate (NAR). This elevated NAR is associated with postoperative complications, prolonged hospital stays, and avoidable healthcare expenditures. Despite international guidelines recommending the routine use of risk prediction models for patients with acute abdominal pain, reported NAR values have reached as high as 28.2% in females and 12.1% in males.

Aim:

The primary study aim is to identify optimal risk prediction models for acute RIF pain in Turkey.

The secondary aims are to audit the normal appendicectomy rate, assess whether these scores have similar efficacy in immigrants, and demonstrate nationwide clinical trends to discuss possible improvements.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients referred to general surgeons with right iliac fossa pain or suspected appendicitis.
* All patients who undergo an appendicectomy during the study period.

Exclusion Criteria:

* Previous appendicectomy, right hemicolectomy, or total colectomy.
* Previous abdominal surgery in the last 90 days.
* Pregnancy.
* Patients confirmed with COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to general surgeons with right iliac fossa pain or suspected appendicitis.
Sampling Method: Non-Probability Sample
Enrollment: 3358 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Best classification performance among 4 appendicitis scoring systems (for Turkish population) | During admission
  Data is used to calculate the four most commonly used adult risk prediction models: Alvarado, the Appendicitis Inflammatory Response (AIR), Raja Isteri Pengiran Anak Saleha Appendicitis (RIPASA), and Adult Appendicitis Score (AAS). Then, the performance of each scoring system will be compared with one another to find the best scoring system among them.

SECONDARY OUTCOMES:
Normal Appendicectomy Rate (NAR) | All patients are followed up for 60 days, and data being utilized for NAR calculation is collected within that timeframe.
  The NAR value is calculated as the percentage of patients with normal appendix histology who had undergone appendectomy. Patients with appendix pathology other than appendicitis (such as appendix tumor) were included in the denominator but not the numerator.
Best classification performance among 4 appendicitis scoring systems (for immigrant population) | During admission
  Data is used to calculate the four most commonly used adult risk prediction models: Alvarado, the Appendicitis Inflammatory Response (AIR), Raja Isteri Pengiran Anak Saleha Appendicitis (RIPASA), and Adult Appendicitis Score (AAS). Then, the performance of each scoring system will be compared with one another to find the best scoring system among them.

CONTACTS AND LOCATIONS:
Overall Officials: Sezai Leventoglu, Professor, Study Chair — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No